CLINICAL TRIAL: NCT04261244
Title: Preoperative Radiotherapy Versus Postoperative Radiotherapy After Neoadjuvant Chemotherapy ("NeoRad") in High-risk Breast Cancer: a Prospektiv, Randomized, International Multicenter Phase III Trial
Brief Title: NeoRad Breast Cancer Study
Acronym: NeoRad
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bielefeld University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeoRad Breast Cancer Study
Record Dates: First submitted 2019-09-30; First posted 2020-02-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: neoadjuvant chemotherapy; preoperative radiotherapy; capsular contraction; immediate reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: randomized, multicenter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): preoperative radiotherapy in breast cancer after neoadjuvant chemotherapy
  Interventions: Radiation: preoperative radiotherapy
- Standard treatment (Active Comparator): standard treatment (postoperative radiotherapy) in breast cancer after neoadjuvant chemotherapy
  Interventions: Radiation: postoperative radiotherapy

INTERVENTIONS:
Radiation: preoperative radiotherapy — preoperative radiotherapy instead of postoperative radiotherapy in breast cancer after neoadjuvant chemotherapy
  Arms: Experimental Arm
Radiation: postoperative radiotherapy — postoperative radiotherapy in breast cancer after neoadjuvant chemotherapy
  Arms: Standard treatment

SUMMARY:
The NEORAD trial tests whether preoperative radiotherapy results in an improved DFS and less radiation induced late effect compared to postoperative radiotherapy in higher risk breast cancer after NACT.

DETAILED DESCRIPTION:
The standard of care for high-risk breast cancer consists of neoadjuvant chemotherapy and surgery followed by postoperative whole breast/chest wall irradiation+/- an additional boost (= irradiation restricted to the tumour bed in the case of breast-conserving therapy). In case of lymph node involvement in most patients require additional radiation of the regional lymph nodes. Adjuvant radiotherapy significantly reduces ipsilateral breast cancer recurrences, breast cancer specific mortality, and overall mortality. The optimal time of radiotherapy in patients, who are candidates for neoadjuvant chemotherapy (NACT) has never been addressed in a randomised controlled trial.

The Study Chairman of the NEORAD trial is Prof. Dr. med. Christiane Matuschek. The deputies of the Study Chairman are Prof. Dr. med. Wilfried Budach and Prof. Dr. med. Tanja Fehm.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive, unilateral breast cancer
* Indication for radiotherapy
* Indication for neoadjuvant chemotherapy (+/- antibody treatment or other targeted therapies) in accordance with national and international guidelines
* Female
* Informed consent for the trial signed by the patient
* Hormone receptor and HER2 status: no restrictions
* All grades G1-G3
* Age ≥ 18 years at the time of informed consent
* Performance status ≤ 2
* No pre-existing conditions that prohibit therapy

Exclusion Criteria:

* Neoadjuvant treatment solely with endocrine therapy
* Bilateral breast cancer
* Pregnancy or lactation
* Prior radiotherapy of the thorax
* Connective tissue disease, including rheumatoid arthritis and thromboangiitis obliterans
* Pre-existing symptomatic chronic lung disease (fibrosis, pneumoconiosis, adult-onset allergies, such as farmer's lung, severe lung emphysema, COPD °III)
* Cardiac comorbidities: symptomatic coronary heart disease, prior heart attack, heart failure NYHA ≥II or AHA ≥C, pacemaker, and/or implanted defibrillator
* Malignoma except basalioma or in-situ-carcinomas in complete response
* Distant metastasis
* Plexopathies of the arm of the treated side
* Stiffness of the shoulder of the arm of the side of the breast cancer of any origin (e.g. following a road accident)
* Lymph edema ≥°II of the arm at the side of the breast cancer
* Other medical conditions that prohibit the neoadjuvant radiotherapy (i.e. Expected non-compliance, etc.)
* Male patients
* Patients who have previously been assessed for chemotherapy response

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1826 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2034-03-31 (Estimated)

PRIMARY OUTCOMES:
disease free survival (DFS): | 6 to 10 years
  Time interval in which the patient does not show any signs or symptoms of the treated cancer (local or regional recurrence, distant metastases, or death of any cause) beginning after randomisation to a study arm.
  This is a way to measure how well the new treatment is working.

SECONDARY OUTCOMES:
local recurrence rate [in affected breast] (LR) | 6 to 10 years
  Rate of cancer that has recurred at the same location as the primary cancer. This is a way to measure how well the new treatment is working.
locoregional recurrence rate (LRR) | 6 to 10 years
  Rate of new cancer at any locations (regional lymph nodes, chest wall/mastectomy site) on side which was previously affected by the primary cancer.
  This is a way to measure how well the new treatment is working.
disease metastases free survival (DMFS) | 6 to 10 years
  Time interval beginning after randomisation in which the patient survives and the cancer has not metastasized.
  This is a way to measure how well the new treatment is working.
overall survival (OS) | 6 to 10 years
  Length of time beginning after randomisation in the study that the patient survives.
  This is a way to measure how well the new treatment is working.
disease specific survival (DSS) | 6 to 10 years
  Length of time from the beginning of the study after randomisation in a study arm that the patient survives the specific cancer.
  This is a way to measure how well the new treatment is working.
Assesment of cosmetic results by the physicians and the patient using a 5 point Scoring System* | 6 to 10 years
  A grading scale is provided for cosmetic results (5 Point Scoring System):
  E0 Excellent aesthetic result: At first sight no visible therapy sequellae. Both breasts have a similar appearance E1 Good: minimal changes in pigmentation, a visible scar, localized teleangieectasia.
  E2 Moderate: marked sequellae with a clear deformation of the breast contour, nipple displacement, or marked skin changes, but yet "acceptable".
  E3 Bad: severe retraction or fibrosis, severe teleangiectasia. E4 Complications: skin necrosis
Assesment of cosmetic results by the physicians using breast retraction assessment-Score (BRA Score)* | 6 to 10 years
  *The BRA Score measures breast symmetry of the treated breast in comparison to the untreated breast. The average in the general population is 1.2 cm. A higher BRA score is worse. A BRA score of 0 cm is optimal.
Measurement of the quality of life (QOL): functional scale | 6 to 10 years
  QoL will be assessed by EORTC (European Organisation for Research and Treatment of Cancer) QLQ-C30 questionnaires for overall QoL and EORTC QLQ-BR23 for breast-specific QoL. The QLQ-C30 consists of 30 questions categorized in functional and symptom-specific scales and provides a global score through two general questions concerning health and quality of life. QLQ-BR23 is a standard instrument for measuring QoL in patients with breast cancer. The questionnaire has 23 items with four possible answers each (not at all, a little, quite a bit, very much). Results are reported using functional scales (e.g. body image, sexual functioning) and symptom-related items (e.g. systemic therapy side effects, breast symptoms). It is also common practice to classify the summary scores into four distinct categories with functional scales (0-25 bad; 26-50 moderate; 51-75 good; 76-100 excellent) and symptom-related scales.
Measurement of the quality of life (QOL): symptom-related scale | 6 to 10 years
  QoL will be assessed by EORTC (European Organisation for Research and Treatment of Cancer) QLQ-C30 questionnaires for overall QoL and EORTC QLQ-BR23 for breast-specific QoL. The QLQ-C30 consists of 30 questions categorized in functional and symptom-specific scales and provides a global score through two general questions concerning health and quality of life. QLQ-BR23 is a standard instrument for measuring QoL in patients with breast cancer. The questionnaire has 23 items with four possible answers each (not at all, a little, quite a bit, very much). Results are reported using functional scales (e.g. body image, sexual functioning) and symptom-related items (e.g. systemic therapy side effects, breast symptoms). It is also common practice to classify the summary scores into four distinct categories with functional scales and symptom-related scales: (0-25 excellent; 26-50 good; 51-75 moderate, 76-100 bad)
Assessment of arm lymphedema rates by the physicians using common toxicity criteria for adverse events CTCAE, version 5.0 | 6 to 10 years
  Lymphedema: 'A disorder characterized by excessive fluid collection in tissues that causes swelling.'
  A grading scale is provided for arm lymphoedema rates higher than Grade 1 of the irradiated side (0= "not present", 1= "Trace thickening or faint discoloration", 2= "Marked discoloration; leathery skin texture; papillary formation; limiting instrumental ADL*", 3= "Severe symptoms; limiting self care ADL") using common toxicity criteria for adverse events CTCAE, version 5.0
  *ADL = activities of daily living
Assessment of plexopathia higher than Grade 1 of brachial plexus on irradiated side by the physicians using common toxicity criteria for adverse events CTCAE, version 5.0 | 6 to 10 years
  Brachial plexopathia:'"A disorder characterized by regional paresthesia of the brachial plexus, marked discomfort and muscle weakness, and limited movement in the arm or hand.'
  A grading scale is provided for plexopathia of brachial plexus on the irradiated side higher than Grade 1 (0= "not present", 1= "Aysmptomatic; clinical or diagnostic observations only; intervention not indicated", 2= "Moderate symptoms; limiting instrumental ADL*", 3= "Severe symptoms, limiting self care ADL") using common toxicity criteria for adverse events CTCAE, version 5.0
  *ADL = activities of daily living
Assessment of treatment-related toxicity measured by the physicians using standardized common toxicity criteria for adverse events CTCAE, version 5.0. | 6 to 10 years
  A grading scale is provided for each side effect (0= not present, 1=asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, 3=moderate; minimal, local or noninvasive intervention indicated; -4=severe or medically significant but not immediately life-threatening)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane M Prof., MD Prof., Study Chair — Bielefeld University
Locations (16):
- Germany (16):
  - St. Marien-Krankenhaus Ahaus, Ahaus
  - Hochtaunus-Kliniken, Bad Homburg
  - Sana Klinikum Lichtenberg, Berlin
  - St. Agnes-Hospital, Bocholt
  - Städtisches Klinikum Dessau, Dessau
  - Universitätsfrauenklinik UK OWL, Klinikum Lippe, Detmold
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Niels-Stensen-Kliniken Franziskus-Hospital Harderberg, Georgsmarienhütte
  - Sana Klinikum Hameln-Pyrmont, Hamelin
  - Sana Klinikum Offenbach, Offenbach
  - medius Klinik Ostfildern-Ruit, Ostfildern
  - Leopoldina Krankenhaus Schweinfurt, Schweinfurt
  - Johanniter-Krankenhaus Stendal, Stendal
  - Rems-Murr-Klinikum Winnenden, Winnenden
  - Helios Universitätsklinikum Wuppertal, Wuppertal
  - Heinrich-Braun-Klinikum, Zwickau

IPD SHARING:
Plan to Share IPD: No